CLINICAL TRIAL: NCT06579677
Title: PRospective Observation on CErebral microvaScular Structure and Function (PROCESS): a Population-based Prospective Cohort Study
Brief Title: PRospective Observation on CErebral microvaScular Structure and Function
Acronym: PROCESS
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Daxing District People Hospital (Unknown)
Responsible Party: Principal Investigator, yilong Wang, Professor, Beijing Tiantan Hospital
Other Study IDs: KY2024-179-02
Record Dates: First submitted 2024-08-23; First posted 2024-08-30 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Microvascular Dysfunction; Cerebral Small Vessel Diseases; Cognitive Dysfunction; Cerebrovascular Disorders; Cardiovascular Diseases; Population
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction; Cerebrovascular Disorders; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples of fasting blood, morning urine, feces, oral plaque bacteria will be collected at baseline to test genetic and metabolomic markers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PROCESS Cohort
  Interventions: Other: Without any intervention

INTERVENTIONS:
Other: Without any intervention — No interventions will be performed.

SUMMARY:
This is a population-based prospective cohort study, aiming to assess the prevalence, distributional characteristics, and dynamic change of cerebral small vessel dysfunction in a Chinese community population using advanced vascular imaging techniques; meanwhile to investigate the effect of vascular risk factors on cerebral small vessel dysfunction, cardiovascular and cerebrovascular diseases, cognitive dysfunction, and mortality.

DETAILED DESCRIPTION:
Brain health is defined as normal brain structure, function and social adaptation and the absence of major brain diseases. Brain health is a lifespan-wide process that can be objectively measured and subjectively perceived and is determined by socio-psycho-biological factors. Currently, neurological disorders are the first cause of healthy life lost and the second leading cause of death globally, with nearly 9 million people dying each year from brain-related diseases.

Prevention of major brain diseases, including stroke and dementia, is first and foremost for brain health management. Notably, cerebral small vessel dysfunction may be an earlier pathologic change for the aforementioned major brain diseases. Cerebral small vessel dysfunction includes increased blood-brain barrier permeability, altered neurovascular coupling, decreased cerebral perfusion, decreased cerebral autoregulation, decreased cerebrovascular reactivity, and altered cerebral resting blood flow. Previous studies have shown that the prevalence of cerebral small vessel dysfunction was as high as 40% to 70% in people with illness but data from the general population remain scarce. Vascular risk factors such as aging, hypertension, diabetes, obesity, dyslipidemia, and insulin resistance have been known as important risk factors for the development of major brain diseases. Whereas, it is unclear whether vascular risk factors will cause these brain diseases through affecting cerebral small vessel function.

Thus, this prospective cohort study aims to assess the prevalence, distributional characteristics, and dynamic change of cerebral small vessel dysfunction, and to investigate the effect of vascular risk factors on cerebral small vessel dysfunction, cardiovascular and cerebrovascular diseases, cognitive dysfunction, and mortality in a Chinese community population.

In this study, a total of 3500 participants aged 50 to 75 years from villages and communities of Daxing District, Beijing will be enrolled using cluster sampling method. All the participants will be interviewed at baseline and followed up for 8 years. Baseline data will be collected through face-to-face interviews by trained interviewers using a standardized questionnaire. Baseline data include demographics, lifestyle, physical activity, medical history, cardiovascular risk factors, dietary habits, medication use, sleep status, novel coronavirus infection. Cognitive function assessment and neuropsychiatric examination will be performed based on various scales such as the Montreal Cognitive Assessment (MoCA) Scale and Mini-Mental State Examination (MMSE) Scale.

Additionally, heart function will be tested using electrocardiogram and color ultrasound. Peripheral vascular examination will be performed to measure ankle-brachial index. Fundus examination will be performed by trained ophthalmologists. Gait and eye movement examination will be performed by trained staff. The body composition will be tested using a body composition analyzer.

The samples of fasting blood, morning urine, feces, oral plaque bacteria will be collected at baseline to test genetic and metabolomic markers. An oral glucose tolerance test will be performed to measure blood glucose, insulin, and C-peptide.

Brain magnetic resonance imaging (MRI) examination will be performed to detect CSVD imaging markers, craniocarotid plaque and stenosis, neurovascular coupling, and cerebral perfusion. The sequences of brain MRI included 3D-T1, 3D-T2, 3D-FLAIR, DWI, HR-MRA, SWI, resting-state fMRI, DTI, ASL, etc. All MRI scans will be conducted on 3.0 T scanners. Imaging data will be saved in digital imaging and communications in medicine (DICOM) format on discs and be analyzed at the Imaging Research Center of Beijing Tiantan Hospital. Transcranial Doppler ultrasonography will be used to detect cerebral autoregulation and cerebral resting blood flow. Carotid ultrasound will be used to measure carotid artery diameter, carotid intramedullary thickness, carotid systolic maximal flow velocity, carotid end-diastolic velocity, pulsatility index, vascular resistance index, carotid artery plaque, carotid artery stenosis, and blood flow velocity.

Routine follow-up will be performed each year to collect cardio-/cerebrovascular diseases and death after enrollment. A further face-to-face interview will be performed at 2, 4, 6, 8 years to collect the data of brain MRI scanning, transcranial Doppler ultrasonography, and cognitive impairment. Meanwhile, standard clinical and neuropsychologic examination will be conducted using the same scale as that at baseline. Fasting blood and morning urine samples will be collected at each follow-up visit following same protocol as that at baseline.

The protocol of this study has been approved by the Ethics Committee of Beijing Tiantan Hospital. All participants will provide written informed consents before entering the study.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling adults aged 50-75 years;
2. Registered Beijing household residents or residents who can be followed up stably in their own communities for a long period;
3. Subjects with written informed consents.

Exclusion Criteria:

1. Residents with moderate to severe disabilities (MRS ≥3), mental illness, stroke, dementia, and other serious neurological disorders (e.g., encephalitis, Parkinson's disease, epilepsy, brain tumors, and rare genetic diseases of the nervous system);
2. Life expectancy of ≤4 years due to serious diseases such as end-stage cancer;
3. Contraindications to magnetic resonance imaging such as implanted devices (e.g., pacemakers, defibrillators, and others);
4. Residents who are participating in other studies.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population of the PROCESS study is community-dwelling adults aged 50-75 years based on cluster sampling from villages and communities of Daxing District, Beijing. The steering committee will attempt to ensure population representativeness of the sample. These selected villages and communities will be living communities (not occupational communities) with little population migration.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2032-03 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Cerebral small vessel disease | 2024-09 to 2032-09
  Cerebral small vessel disease will be evaluated using 3.0 T MRI based on imaging markers of asymptomatic cerebral infarction, cerebral microbleeds, lacunar, white matter hyperintensity, enlarged perivascular space, and cerebral atrophy.
Neurovascular coupling | 2024-09 to 2032-09
  Neurovascular coupling is one of cerebral small vessel function indicators and will be measured by 3.0 T MRI.
Cerebral perfusion | 2024-09 to 2032-09
  Cerebral perfusion is one of cerebral small vessel function indicators and will be measured by 3.0 T MRI.
Cerebral autoregulation | 2024-09 to 2032-09
  Cerebral autoregulation is one of cerebral small vessel function indicators and will be measured by transcranial Doppler ultrasonography.
Cerebral resting blood flow | 2024-09 to 2032-09
  Cerebral resting blood flow is one of cerebral small vessel function indicators and will be measured by transcranial Doppler ultrasonography.

SECONDARY OUTCOMES:
Composite vascular events | 2024-09 to 2032-09
  Composite vascular events include non-fatal acute myocardial infarction, non-fatal acute stroke (cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage), hospitalization for vascular reasons (including unstable angina pectoris, transient ischemic attack, and other ischemic vascular events), and vascular deaths (fatal infarcts, fatal strokes, and other vascular deaths). These events will be collected by self-report and confirmed by reviewing their medical records.
Cognitive impairment measured by the Montreal Cognitive Assessment (MoCA) scale | 2024-09 to 2032-09
Cognitive impairment measured by the Mini-Mental State Examination (MMSE) scale | 2024-09 to 2032-09
All causes of death | 2024-09 to 2032-09
  All causes of death includes cardiovascular death and noncardiovascular death.
Atherosclerotic plaque in retinal arteries. | 2024-09 to 2032-09
Atherosclerotic plaque in craniocarotid arteries. | 2024-09 to 2032-09
Other vascular events | 2024-09 to 2032-09
  Other vascular events include peripheral vascular disease, subclavian steal syndrome and systemic thromboembolic events.
Vascular interventions | 2024-09 to 2032-09
  Vascular interventions such as arterial bypass, balloon dilatation, stent implantation, carotid endarterectomy, mechanical thrombolysis and ischemic amputation. These events will be collected by self-report and confirmed by reviewing their medical records.
Mean blood flow velocity in arteries | 2024-09 to 2032-09
  Mean blood flow velocities in the distal common carotid artery, internal carotid artery bulb, proximal-distal internal carotid artery, and vertebral artery will be measured by pulsed Doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing, Beijing Municipality
  - Beijing Daxing District People Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
The data can be requested through the website of the data management system (http://paper.ncrcnd.org.cn/) or by sending email to the principal investigators.